CLINICAL TRIAL: NCT02503527
Title: Effects of a Diabetes-specific Tube Feed on Glycemic Variability in Critically Ill Patients During Insulin Blood Glucose Management
Brief Title: Efficacy and Safety Study of a Low-carbohydrate Tube Feed in Critically Ill Patients Under Insulin Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low Recruitment rate
Sponsor: Fresenius Kabi (Industry)
Collaborators: OE Clinical Trial Center (KKS) Universität Innsbruck (Unknown); International Medical Research - Partner GmbH (Other); dsh statistical services GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DBHP-001-CEN
Record Dates: First submitted 2015-07-10; First posted 2015-07-21 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: Enteral nutrition; Tube feeding; Diet, carbohydrate-restricted; Diabetes; Aneurysmal Subarachnoid Hemorrhage; Blood glucose; Insulin
MeSH Terms: conditions — Subarachnoid Hemorrhage; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diben 1.5 kcal HP (Other): Diben 1.5 kcal HP, Food for Special Medical Purposes (diabetes-specific tube feed)
  Interventions: Other: Diben 1.5 kcal HP
- Fresubin HP Energy Fibre (1.5 kcal) (Other): Fresubin HP Energy Fibre (1.5 kcal), Food for Special Medical Purposes (standard tube feed)
  Interventions: Other: Fresubin HP Energy Fibre (1.5 kcal)

INTERVENTIONS:
Other: Diben 1.5 kcal HP — Continuous (24h) application according to a standardized enteral feeding protocol via nasogastric tube or percutaneous endoscopic gastrostomy (PEG); pump-assisted application (Charriére (CH) > 8), duration according to patient's tolerance and requirements for a maximum of 5 days. Dosage: 21 - 24 kcal/kg body weight/day (corresponding to 14 to 16 ml/kg body weight/day).
  Arms: Diben 1.5 kcal HP
Other: Fresubin HP Energy Fibre (1.5 kcal) — Continuous (24h) application according to a standardized enteral feeding protocol via nasogastric tube or percutaneous endoscopic gastrostomy (PEG); pump-assisted application (Charriére (CH) > 8), duration according to patient's tolerance and requirements for a maximum of 5 days. Dosage: 21 - 24 kcal/kg body weight/day (corresponding to 14 to 16 ml/kg body weight/day).
  Arms: Fresubin HP Energy Fibre (1.5 kcal)

SUMMARY:
The purpose of this study is to determine the efficacy and safety of a diabetes-specific tube feed in comparison to an isocaloric, isonitrogenous standard enteral formula in critically ill patients receiving insulin treatment for blood glucose management.

ELIGIBILITY:
Inclusion Criteria:

* Patients with spontaneous aneurysmal subarachnoid hemorrhage (SAH) defined according to Hunt and Hess scale grade HH5
* Requiring mechanical ventilation in the ICU at the time of enrolment
* Enteral nutrition (EN) in the ICU at time of enrolment

  * If enrolment on day 3 of ICU stay, EN equal to or larger than 80% of total calories in case of supplementary parenteral nutrition (PN) with anticipated 100% EN as of day 4 to 8 of ICU stay
  * If enrolment on day 4 of ICU stay, 100% EN planned for at least 5 days from the time of enrolment
* Patients expected to stay in the ICU for at least 5 days following enrolment
* Age 18 - 75 years
* Glycemic control with intravenous insulin therapy to maintain a target glucose range between 110 mg/dL and 150 mg/dL (6.1 and 8.3 mmol/l)
* Informed consent according to local regulations for decisionally impaired subjects

Exclusion Criteria:

* Patients with septic shock at time of enrolment
* Participation in a clinical trial with any investigational product within 4 weeks before study
* Patients requiring a fibre free diet
* Total or supplementary parenteral nutrition (> 20% of total calories)
* Known or suspected intolerance or allergy to any component of the study product(s), e.g. galactosemia
* Gastrectomy
* Postpyloric nutrition
* Any clinical condition not allowing enteral nutrition (e.g. emesis, severe reflux, severe diarrhea)
* Known severe heart failure (NYHA class 4)
* Liver insufficiency / failure (male: ALAT > 150 U/l; female: ALAT > 120 U/l)
* Acute kidney failure (blood creatinine > 2.5 mg/dl)
* Body Mass Index < 18 or > 35 kg/m²
* Known or suspicion of drug abuse
* Pregnant or breast feeding women
* Patients with diabetes mellitus type I

Exclusion After Enrolment (Withdrawal of Subjects)

* Start of PN with more than 20% of total given energy amount/ day
* Insulin infusion stopped unexpectedly for > 12h for non-nutritional reasons
* Discharge from ICU
* Intolerable AEs
* Major protocol violation
* Withdrawal of informed consent
* Discontinuation of study treatment for other reasons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-08; Primary Completion 2018-08 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Blood glucose variability (within patient standard deviation of blood glucose values per day) | At Day 3 of intervention or the day prior to switch from intravenous to subcutaneous insulin administration, whichever comes first

SECONDARY OUTCOMES:
Glucose variability | Days 2, 4 and 5 of intervention
Time to switch from intravenous to subcutaneous insulin administration | Days 1-6, daily
Insulin requirements in IU per day | Days 1 - 6, daily
Blood glucose levels | Days 1 - 6, daily
HbA1c | Days 1, 6, 28
Difference between target and given enteral nutrition (Compliance) | Days 2-6, daily
Cerebral and subcutaneous microdialysis: glucose | Days 1 - 6, daily
Cerebral and subcutaneous microdialysis: lactate/pyruvate ratio | Days 1 - 6, daily
Hospital mortality | Day 28
ICU mortality | Day 28
ICU length of stay | Day 28
Days of mechanical ventilation | Day 28
Non-gastrointestinal complications (AEs) to enteral nutrition and application | Days 2-6, daily
Gastro-intestinal intolerance (AEs, complications) | Days 2-6, daily

CONTACTS AND LOCATIONS:
Overall Officials: Ronny Beer, PD Dr. med., Principal Investigator — Medical University of Innsbruck, Department of Neurology, Neurocritical Care Unit
Locations (1):
- Universitätsklinikum Innsbruck, Innsbruck, Austria